CLINICAL TRIAL: NCT02861781
Title: Study of New Determinants of Type 2 Diabetes in Severe Obesity
Brief Title: Collection of Human Metabolic Tissues
Acronym: COMET
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL15_0271; 2015-A01193-46 (Other: French Agency for the Safety of Health Products); UF 9605 (Other: Montpellier University Hospital)
Record Dates: First submitted 2016-08-02; First posted 2016-08-10 (Estimated); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Obesity; Insulin Resistance; Diabetes Mellitus, Type 2
Keywords: Bariatric surgery
MeSH Terms: conditions — Obesity; Insulin Resistance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Type 2 diabetes: Type 2 diabetes according to ADA criteria
  Interventions: Other: Collection of blood samples and tissues
- Insulin resistance non diabetes: HOMA-IR criteria ≥ 3
  Interventions: Other: Collection of blood samples and tissues
- Insulin sensitivity non diabetes: HOMA-IR criteria < 3
  Interventions: Other: Collection of blood samples and tissues

INTERVENTIONS:
Other: Collection of blood samples and tissues — Collection of blood samples and tissues during bariatric surgery and blood samples during followup visits

SUMMARY:
This project aims at identifying new determinants of type 2 diabetes in severe obesity. To do so, a biological collection, including tissues of interest in the field of metabolism, will be collected during bariatric surgery in obese patients. Three different groups of metabolic status of patients, corresponding to different stages of evolution of the disease, will be constituted: type 2 diabetes, insulin resistance, insulin sensitivity.

The main objective is to compare, between these 3 groups of patients, several biological processes that may be involved in the pathophysiology of type 2 diabetes and disorders associated with obesity, including:

* Abnormalities of the transcriptome, proteome, metabolome in all target tissues (plasma, serum, muscle, subcutaneous and visceral adipose tissue, omental artery, liver)
* Identification of metabolic signatures, protein and miRNA in plasma
* Immunoinflammatory response in adipose tissue
* Polymorphisms SNP from whole blood
* Histological analysis of tissue sections This main objective will be studied on samples taken at the time of surgery Secondary objectives will be to study the changes in metabolites, proteins and miRNA in plasma level 3 and 12 months after the completion of surgery, according to the initial metabolic state.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Age 18 - 65 years inclusive at surgery
3. IMC > 35
4. Subject qualified for bariatric surgery (sleeve gastrectomy or gastric bypass)
5. Specific criteria :

   * Type 2 diabetes group (D) (90 patients) : type 2 diabetes according to ADA criteria
   * Insulin resistance non diabetes group (IR) (80 patients) : HOMA-IR criteria ≥ 3
   * Insulin Sensitivity non diabetes group (N) (100 patients) : N1.HOMA-IR criteria < 3

Non inclusion Criteria:

1. Vulnerability according to article L1121-6 of the Public Health Code
2. Protected adult or unability to give consent according to article L1121-8 of the Public Health Code
3. Unability to understand the design and aims of the study or to communicate with the investigator
4. Non affiliation to a social security system
5. Prior bariatric surgery (except lap-band procedure)
6. Serologic profile indicating hepatitis B, hepatitis C or HIV infection
7. Inflammatory, infectious or autoimmune disease (current or in the previous 3 month)
8. Malignancies within 5 years prior to inclusion or not considered as treated curatively
9. Concomitant use of steroids or NSAI or use in the 8 days before surgery
10. alcohol abuse/addiction
11. Anticipated poor compliance to study procedures
12. Other type of diabetes than type 2

Exclusion Criteria :

1. Cancelled bariatric surgery
2. Tissue collection not possible during the bariatric surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject qualified for bariatric surgery
Sampling Method: Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2016-02-02 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
comparison of metabolites | At baseline (day of surgery)
comparison of proteins levels | At baseline (day of surgery)
  in liver, muscle, adipose tissue and plasma according to metabolic state
comparison of miRNA | At baseline (day of surgery)
  in liver, muscle, adipose tissue and plasma according to metabolic state

SECONDARY OUTCOMES:
changes in metabolites in plasma level | 3 and 12 months after the completion of surgery
changes in proteins in plasma level | 3 and 12 months after the completion of surgery
changes in miRNA in plasma level | 3 and 12 months after the completion of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Florence GALTIER, Principal Investigator — Montpellier University Hospital
Locations (1):
- Hôpital Saint Eloi, Montpellier, France